CLINICAL TRIAL: NCT07073950
Title: A Randomised, Double-blind, Multi-centre, Placebo-controlled, Crossover Study to Assess the Effect of Budesonide/Glycopyrronium/Formoterol Fumarate Metered Dose Inhaler on Cardiac and Lung Function in Participants With Chronic Obstructive Pulmonary Disease and Hyperinflation
Brief Title: A Study to Investigate the Effect of Budesonide/Glycopyrronium/Formoterol Fumarate Metered Dose Inhaler (BGF MDI) Compared With Placebo MDI on Heart and Lung Function in Participants With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: ORATOS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D5980C00048; 2025-521987-37-00 (Other: EU CT Number)
Record Dates: First submitted 2025-07-17; First posted 2025-07-20 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hyperinflation
Keywords: Metered Dose Inhalers (MDI); Inhaled Corticosteroid (ICS); Long-acting muscarinic antagonist (LAMA); Long-acting beta2 agonist (LABA)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Sequence 1: BGF MDI and Placebo (Experimental): Participants will receive BGF MDI in Period 1 followed by Placebo in Period 2.
  Interventions: Drug: Budesonide/Glycopyrronium/Formoterol Fumarate; Drug: Placebo; Device: Metered dose inhaler
- Sequence 2: Placebo and BGF MDI (Experimental): Participants will receive Placebo in Period 1 followed by BGF MDI in Period 2.
  Interventions: Drug: Budesonide/Glycopyrronium/Formoterol Fumarate; Drug: Placebo; Device: Metered dose inhaler

INTERVENTIONS:
Drug: Budesonide/Glycopyrronium/Formoterol Fumarate — BGF will be administered as 2 inhalations via oral route of administration
Drug: Placebo — Matching placebo will be administered as 2 inhalations via oral route of administration
Device: Metered dose inhaler — Participants will receive BGF and matching placebo via metered dose inhaler in treatment periods of the study.

SUMMARY:
The purpose of the study is to evaluate the effect of BGF MDI compared with placebo MDI on cardiac and lung function when administered in participants diagnosed with COPD and hyperinflation.

DETAILED DESCRIPTION:
This is a Phase IV, randomised, double blind, multiple centre, placebo controlled, crossover study where the effectiveness of BGF MDI in comparison with matching placebo MDI on cardiac and pulmonary function will be evaluated in patients with COPD and hyperinflation.

The study will comprise of:

* Screening period
* Participants will receive placebo inhaler and salbutamol before randomization
* Two treatment periods where participants will be randomized 1:1 to receive either the study intervention BGF MDI followed by matching placebo or study interventions in reverse order
* A final follow-up period

ELIGIBILITY:
Key Inclusion Criteria:

* Current or former smoker with a history of ≥ 10 pack-years of tobacco smoking.
* A diagnosis of COPD confirmed by a post-bronchodilator forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) < 0.7.
* At Visit 1: A pre-bronchodilator FEV1 < 80%.
* At Visit 1: Peripheral blood eosinophil count < 300 cells/cubic millimeter (mm³), with no recorded history of eosinophil count > 300 cells/mm³ in the past 12 months.
* At Visit 1: Modified Medical Research Council (mMRC) ≥ 1.
* At Visit 2: A pre-bronchodilator functional residual capacity (FRC) of > 135% of predicted normal FRC.
* At Visit 2: A post-bronchodilator FEV1 ≥ 30% and < 80% of the predicted normal value.
* Participants must be on mono-, dual-, or triple-inhaled maintenance COPD treatment.
* Female participants must either be not of childbearing potential or using a form of highly effective birth control.
* All women of child bearing potential must have a negative pregnancy test at the Visit 1.

Exclusion Criteria:

* A current diagnosis of asthma, asthma-COPD overlap, or any other chronic respiratory disease other than COPD, such as alpha-1 antitrypsin deficiency, active tuberculosis, lung cancer, lung fibrosis, sarcoidosis, interstitial lung disease, and pulmonary hypertension.
* History of a COPD exacerbation that required hospitalisation, or 2 or more COPD exacerbations that required systemic corticosteroids.
* History of myocardial infarction or acute coronary syndrome.
* History or current atrial or ventricular arrhythmia to be confirmed by electrocardiogram (ECG).
* Participants with a cardiac implantable electronic device, including pacemaker, implantable cardioverter defibrillator, or cardiac resynchronization therapy.
* Participants with ECG QTcF interval at Visit 1 > 460 milliseconds (ms) for males and > 480 ms for females.
* Participants who have had a respiratory tract infection within 8 weeks prior to Visit 1 and/or during the screening/run-in period.
* Participants with lung lobectomy, lung volume reduction (during the study and within 3 months of Visit 1), or lung transplantation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in left ventricular end diastolic volume (LVEDV) measured by magnetic resonance imaging (MRI) | Up to 3 weeks
  The effect of BGF relative to placebo on LVEDV in participants with COPD and hyperinflation will be evaluated.

SECONDARY OUTCOMES:
Change from baseline in functional residual capacity/total lung capacity (FRC/TLC) measured by body plethysmography | Up to 3 weeks
  The effect of BGF relative to placebo on FRC/TLC will be evaluated.
Change from baseline in residual volume/total lung capacity (RV/TLC) measured by body plethysmography | Up to 3 weeks
  The effect of BGF relative to placebo on RV/TLC will be evaluated.

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (3):
  - Research Site, Ahrensburg
  - Research Site, Berlin
  - Research Site, Hanover
- United Kingdom (3):
  - Research Site, Harefield
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secureresearchenvironmentVivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/